CLINICAL TRIAL: NCT02952014
Title: Pharmacokinetic, Thermogenic, Hemodynamic, Ergogenic Assessment of a Pre-Workout Dietary Supplement
Brief Title: Assessment of a Pre-Workout Dietary Supplement
Acronym: NB1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrabolt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2014-0022FX
Record Dates: First submitted 2016-09-13; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C4 Extreme (Experimental): One dose of 12 grams (powder mixed with water): 1500 mg beta alanine, 1000 mg creatine nitrate, 1000 mg arginine AKG, 250 mg vitamin C, 150 mg n-acetyle tyrosine, 135 mg caffeine, 7.5 mg l-dopa, 30 mg vitamin B3, 10 mg synephrine, 0.5 mg vitamin B6, 0.25 mg vitamin B9, 0.035 mg vitamin B12.
  Interventions: Dietary Supplement: C4 Extreme
- C4 Extreme (without Advantra Z) (Active Comparator): One dose of 12 grams (powder mixed with water): 1500 mg beta alanine, 1000 mg creatine nitrate, 1000 mg arginine AKG, 250 mg vitamin C, 150 mg n-acetyle tyrosine, 135 mg caffeine, 7.5 mg l-dopa, 30 mg vitamin B3, 0.5 mg vitamin B6, 0.25 mg vitamin B9, 0.035 mg vitamin B12.
  Interventions: Dietary Supplement: C4 Extreme (without Advantra Z
- Placebo (Placebo Comparator): One dose of flavored placebo (powder mixed with water)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: C4 Extreme — Pre-Workout Dietary Supplement
  Arms: C4 Extreme
Dietary Supplement: C4 Extreme (without Advantra Z — Pre-Workout Dietary Supplement
  Arms: C4 Extreme (without Advantra Z)
Dietary Supplement: Placebo — Pre-Workout Dietary Supplement
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the acute effects of a pre-workout dietary supplement on energy metabolism, cardiovascular hemodynamics, blood metabolites and mental focus.

DETAILED DESCRIPTION:
A number of nutritional strategies have been developed to optimize nutrient delivery prior to exercise. This includes providing carbohydrate and a number of ergogenic nutrients prior to, during and/or following exercise. As a result a number of pre-workout supplements have been developed to increase energy availability, promote vasodilation and/or positively affect exercise capacity. The purpose of this study is to investigate the potential ergogenic value of acute ingestion of a pre-workout dietary supplement prior to exercise.

ELIGIBILITY:
Inclusion Criteria:

* you are an apparently healthy and recreationally active man or woman between the ages of 18 and 40;
* you will need to have at least six months immediate prior history of resistance training on the bench press and leg press or squat;

Exclusion Criteria:

* you have a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypo-tension, thyroid disease, arrhythmia and/or cardiovascular disease;
* you are currently using prescription medications;
* you have an intolerance to caffeine and/or other natural stimulants;
* you are pregnant or a lactating female or plan to become pregnant with the next month;
* you have a history of smoking;
* you drink excessively (i.e., 12 drinks per week or more);

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Optimize nutrient delivery prior to exercise by assessing; cognitive function (i.e., Stroop Color and Word Test and Word Recall Test). | Three weeks
Optimize nutrient delivery prior to exercise by assessing Readiness to Perform Visual Analog Scale. | Three weeks
Optimize nutrient delivery prior to exercise by assessing Resting Energy Expenditure. | Three weeks
Optimize nutrient delivery prior to exercise by assessing Heart Rate. | Three weeks
Optimize nutrient delivery prior to exercise by assessing Blood Pressure. | Three weeks
Optimize nutrient delivery prior to exercise by assessing ECG. | Three weeks

SECONDARY OUTCOMES:
Measure standard clinical chemistry panels in the blood to evaluate safety. | Three weeks
Measure Heart Rate to evaluate safety. | Three weeks
Measure Blood Pressure to evaluate safety. | Three weeks
Measure ECG to evaluate safety. | Three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Laboratory, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung YP, Earnest CP, Koozehchian M, Galvan E, Dalton R, Walker D, Rasmussen C, Murano PS, Greenwood M, Kreider RB. Effects of acute ingestion of a pre-workout dietary supplement with and without p-synephrine on resting energy expenditure, cognitive function and exercise performance. J Int Soc Sports Nutr. 2017 Jan 12;14:3. doi: 10.1186/s12970-016-0159-2. eCollection 2017. PMID 28096758